CLINICAL TRIAL: NCT06232200
Title: Investigation of the Effectiveness of Acupuncture in Patients Diagnosed With Interstitial Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ali Ihsan Memmi, Medical Doctor, Medipol University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34043404
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-02

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: acupuncture; Interstitial Cystitis; Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The conventional treatment group will be determined as the control group and the patients in the treatment group will receive acupuncture treatment twice a week, a total of 8 sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL GROUP (No Intervention): REGULAR TREATMENT
- ACUPUNCTUR GROUP (Experimental): Acupuncture application will be performed by bilateral needling of The Sanyinjiao (SP6), Yin Ling Quan (SP9), Zu San Li, "Leg Three Mile" (ST36) , Tai Chong (LIV3), Hegu (LI4), Taixi (KID3) , Zhongliao (BL33) and Guan Yuan (CV4) acupuncture points using sterile, disposable metal acupuncture needles. The needles will remain in place for approximately 20 minutes during the treatment, a total of 8 sessions are planned, 2 per week.
  Interventions: Other: ACUPUNCTURE

INTERVENTIONS:
Other: ACUPUNCTURE — Acupuncture application will be performed by bilateral needling of The Sanyinjiao (SP6), Yin Ling Quan (SP9), Zu San Li, "Leg Three Mile" (ST36) , Tai Chong (LIV3), Hegu (LI4), Taixi (KID3) , Zhongliao (BL33) and Guan Yuan (CV4) acupuncture points using sterile, disposable metal acupuncture needles. The needles will remain in place for approximately 20 minutes during the treatment, a total of 8 sessions are planned, 2 per week.
  Arms: ACUPUNCTUR GROUP

SUMMARY:
Interstitial cystitis/bladder pain syndrome is a non-bacterial chronic inflammatory disease of the bladder characterized by lower urinary tract symptoms such as dysuria, irritating urgency, and nocturia, as well as pelvic pain associated with bladder filling.

The International Continence Society (ICS) defines bladder pain syndrome as "a complaint of suprapubic pain due to bladder filling accompanied by urinary system symptoms such as increased daytime and nighttime urinary frequency as a result of the exclusion of proven urinary infection or other obvious pathologies." Acupuncture is an important treatment method of traditional Chinese medicine that has been used for more than 2500 years and is performed by placing needles at specific points on the skin.

In the literature, clinical studies have been conducted to evaluate the effectiveness of acupuncture in Interstitial Cystitis and its effectiveness in relieving symptoms has been demonstrated. In the light of these data, our aim in our multi-centered study is to investigate the effectiveness of acupuncture in relieving symptoms and improving the quality of life in patients diagnosed with Interstitial Cystitis.

In our study, patients who applied to the Urology Clinic between 01.02.2024 and 01.07.2024 with pelvic pain or discomfort lasting more than 6 months and lower urinary tract symptoms such as frequent urination, dysuria and nocturia will be examined and evaluated with suspicion of Interstitial Cystitis diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* who diagnosed IC/BPS
* between 30-65 years old
* female

Exclusion Criteria:

* Patients who do not meet the IC/BPS diagnostic criteria,
* who have previously received acupuncture treatment,
* who have localized skin infections involving the acupuncture areas,
* who have bleeding diathesis and who use anticoagulant drugs,
* who cannot comply with the treatment and follow-up schedule will not be included in the study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
O'Leary-Saint symptom score | 1. 6. ve 12. month
  The O'Leary-Saint symptom score is also known as the Interstitial Cystitis Symptom Index and Interstitial Cystitis Problem Index (ICPI). That assesses the 4 core symptoms of Interstitial Cystitis (bladder pain, urgency, frequent urination, and nocturia) by asking the patient how often each is experienced. In this evaluation, the patient is asked to rate the 4 basic symptoms in the Interstitial Cystitis Symptom Index from 0 to 5, according to the patient's complaint, and the 4 basic problems in the Interstitial Cystitis Problem Index from 0 to 4.The goal of this instrument is to evaluate and diagnose patients with IC. The O'Leary-Sant instrument is comprised of a Symptom Index (score range: 0-20 points) and a Problem Index (score range: 0-16 points), each of which contains four questions related to urinary and pain symptoms. For each index, the score is calculated by summing the points for each item. On either index, a score ≥6 points indicates Interstitial Cystitis.

CONTACTS AND LOCATIONS:
Locations (1):
- istanbul Çam Sakura city hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sonmez MG, Kozanhan B. Complete response to acupuncture therapy in female patients with refractory interstitial cystitis/bladder pain syndrome. Ginekol Pol. 2017;88(2):61-67. doi: 10.5603/GP.a2017.0013. PMID 28326514